CLINICAL TRIAL: NCT01755117
Title: Comparison of Posterior Lumbar Plexus Block Plus Sciatic Nerve Block With Sciatic Plus Femoral Plus Obturator Nerve Block for Total Knee Replacement (TKR)
Brief Title: Ultrasound Guided Obturator Nerve Block for Total Knee Replacement (TKR)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Larissa University Hospital (Other)
Responsible Party: Principal Investigator, Marina Simaioforidou, Anesthesiologist, Larissa University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: TKR obturator
Record Dates: First submitted 2012-12-18; First posted 2012-12-24 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Total Knee Replacement; Surgery
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TKR, sciatic, femoral, obturator (Active Comparator): TKR surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block
  Interventions: Other: Sciatic, femoral, obturator nerve blocks
- TKR sciatic nerve block, posterior lumbar plexus block (Active Comparator): TKR surgery under ultrasound guided sciatic nerve block plus posterior lumbar plexus block
  Interventions: Other: Sciatic nerve block, posterior lumbar plexus block

INTERVENTIONS:
Other: Sciatic, femoral, obturator nerve blocks
  Other Names: Ultrasound guided blocks with ropivacaine
  Arms: TKR, sciatic, femoral, obturator
Other: Sciatic nerve block, posterior lumbar plexus block
  Other Names: Ultrasound guided blocks with ropivacaine
  Arms: TKR sciatic nerve block, posterior lumbar plexus block

SUMMARY:
Total Knee Replacement can be performed under the combination of posterior lumbar plexus block plus sciatic nerve block. The investigators can have the same outcome by performing instead of posterior lumbar plexus block more peripheral nerve blocks. More specifically under the combination of sciatic nerve block plus femoral nerve block plus obturator nerve block.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 yrs
* ASA I - III
* TKR surgery

Exclusion Criteria:

* Coagulopathy disorders
* Infection at the puncture site for the interscalene block
* Neurologic deficit in the arm that is going to be operated
* Allergy to local anesthetics
* BMI > 35
* Psychiatric disorders
* Patient's refusal
* Problems with patient communication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Feasibility of TKR surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block measured with Pain Score on the Visual Analog Scale | Completion of surgery
  If the patient complains for pain > 4 in VAS and there is no relief with fentanyl administration the anesthesia plan converts to general anesthesia with laryngeal mask

SECONDARY OUTCOMES:
Intraoperative opioid consumption for TKR surgery under ultrasound guided sciatic nerve block plus femoral nerve block plus obturator nerve block | Intaoperatively

OTHER OUTCOMES:
Postoperative opioid consumption | First 24 postoperative hours

CONTACTS AND LOCATIONS:
Overall Officials: Marina Simaioforidou, Medicine, Principal Investigator — Larissa University Hospital; Metaxia Bareka, Medicine, Study Chair — Larissa University Hospital; George Basdekis, Medicine, Study Chair — Larissa University Hospital; Athanasios Drakos, Medicine, Study Chair — Larissa University Hospital; Aristeidis Zibis, Medicine, Study Chair — Private Clinic of Larissa Asklipeiio; Konstantinos Alexiou, Medicine, Study Chair — Larissa University Hospital
Locations (1):
- Larissa University Hospital, Larissa, Thessally, Greece

REFERENCES:
- [Background] Enneking FK, Chan V, Greger J, Hadzic A, Lang SA, Horlocker TT. Lower-extremity peripheral nerve blockade: essentials of our current understanding. Reg Anesth Pain Med. 2005 Jan-Feb;30(1):4-35. doi: 10.1016/j.rapm.2004.10.002. No abstract available. PMID 15690265